CLINICAL TRIAL: NCT02163642
Title: Bronchial Infections in Patients With Non-Cystic Fibrosis (CF) Bronchiectasis; Role of Innate Lung Defense Mechanisms and Utility of an Electronic Nose for Its Diagnosis
Brief Title: Role of Innate Immunity in Non-Cystic Fibrosis Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-BRO-2013-154
Record Dates: First submitted 2014-05-19; First posted 2014-06-13 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Immunity
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Serum samples
  * Sputum samples and cultures
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-CF Bronchiectasis: Cyranose® 320
  Interventions: Device: Cyranose® 320

INTERVENTIONS:
Device: Cyranose® 320 — Detection of patterns of specific Volatile Organic Compounds in exhaled air

SUMMARY:
The purpose of this study is to demonstrate that 1) the secretion of mucins, antimicrobial peptides and Toll-like receptors is altered in certain patients with non-CF bronchiectasis, which makes them more susceptible to be infected by potentially pathogenic bacteria (PPB); and 2) the electronic nose is able to detect patterns of specific Volatile Organic Compounds (VOC) for patients with non-CF bronchiectasis colonized by PPB.

DETAILED DESCRIPTION:
Prospective, observational study, which will include 50 patients with non-CF bronchiectasis who will be followed for a period of 12 months. A follow up control will be performed every three months to all patients, consisting in medical record, lung function tests, blood and serum collection, sputum analysis and culture, and collection of exhaled air for analysis using an electronic nose. These tests will also be repeated whenever the patient has an exacerbation. At the beginning and end of the study, a high resolution chest CT will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non- CF bronchiectasis based on at least 1 lobe with bronchial dilatation and compatible clinical symptoms such as cough, sputum production and respiratory infections.
* Signed informed consent.

Exclusion Criteria:

* Presence of exacerbation in the last 4 weeks.
* Antibiotic treatment in the last 4 weeks
* Use of oral corticosteroids in the last 4 weeks
* Concomitant terminal illness.
* Current cigarette smoking
* Active allergic bronchopulmonary aspergillosis
* Diagnosis of tuberculosis or active non-tuberculous Mycobacterial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of non-CF bronchiectasis will be recruited from the outpatient clinic of the Pneumology Service of the Sant Pau Hospital in Barcelona
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in sputum mucin levels at 12 months | Baseline and 12 months
  Mucin levels in sputum will be determined with ELISA kits

SECONDARY OUTCOMES:
Change from baseline in sputum mucin levels at 3 months | Baseline and 3 months
  Mucin levels in sputum will be determined with ELISA kits
Change from baseline in sputum mucin levels at 6 months | Baseline and 6 months
  Mucin levels in sputum will be determined with ELISA kits
Change from baseline in sputum mucin levels at 9 months | Baseline and 9 months
  Mucin levels in sputum will be determined with ELISA kits

OTHER OUTCOMES:
Change from baseline in patterns of specific volatile organic compounds in exhaled air at 3 months | Baseline and 3 months
  The patterns of specific volatile organic compounds in exhaled air will be determined with the electronic nose device (Cyranose® 320).
Change from baseline in patterns of specific volatile organic compounds in exhaled air at 6 months | Baseline and 6 months
  The patterns of specific volatile organic compounds in exhaled air will be determined with the electronic nose device (Cyranose® 320).
Change from baseline in patterns of specific volatile organic compounds in exhaled air at 9 months | Baseline and 9 months
  The patterns of specific volatile organic compounds in exhaled air will be determined with the electronic nose device (Cyranose® 320).
Change from baseline in patterns of specific volatile organic compounds in exhaled air at 12 months | Baseline and 12 months
  The patterns of specific volatile organic compounds in exhaled air will be determined with the electronic nose device (Cyranose® 320).

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Sibila, MD PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain